CLINICAL TRIAL: NCT01947140
Title: Phase I/IIA Study of the Novel Antifolate Agent Pralatrexate in Combination With the Histone Deacetylase Inhibitor Romidepsin for the Treatment of Patients With Peripheral T-cell Lymphoma
Brief Title: Pralatrexate + Romidepsin in Relapsed/Refractory Lymphoid Malignancies
Acronym: PDX+Romi
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jennifer Amengual (Other)
Responsible Party: Sponsor-Investigator, Jennifer Amengual, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ5656
Record Dates: First submitted 2013-09-09; First posted 2013-09-20 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Lymphoid Malignancies; Multiple Myeloma; Lymphoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: Lymphoid Malignancies; Multiple Myeloma; Lymphoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma; Follicular Lymphoma; Diffuse Large B-Cell Lymphoma; Anaplastic Large Cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — 10-propargyl-10-deazaaminopterin; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I: Schedule A (Experimental): Subjects will receive dose escalation of pralatrexate and romidepsin, receiving both infusions on days 1 and 8 of each 21 day cycle
  Interventions: Drug: Pralatrexate; Drug: Romidepsin
- Phase I: Schedule B (Experimental): Subjects will receive dose escalation of pralatrexate and romidepsin, receiving both infusions on days 1 and 15 of each 28 day cycle
  Interventions: Drug: Pralatrexate; Drug: Romidepsin
- Phase II (Experimental): Subjects will receive Pralatrexate 25 mg/m2 and Romidepsin 12 mg/m2 will be given intravenously once weekly on days 1 and 15 on a 28 day cycle
  Interventions: Drug: Pralatrexate; Drug: Romidepsin

INTERVENTIONS:
Drug: Pralatrexate — Phase I - Schedule A: Intravenous drug given on days 1 and 8 of each 21 day cycle Schedule B: Intravenous drug given on days 1 and 15 of each 28 day cycle Dose escalation from 10 mg/m2 to 25 mg/m2
  Phase II - 25 mg/m2 will be given intravenously once weekly on days 1 and 15 on a 28 day cycle.
  Other Names: Folotyn
Drug: Romidepsin — Phase I - Schedule A: Intravenous drug given on days 1 and 8 of each 21 day cycle Schedule B: Intravenous drug given on days 1 and 15 of each 28 day cycle Dose escalation from 12 mg/m2 to 14 mg/m2.
  Phase II - 12 mg/m2 will be given intravenously once weekly on days 1 and 15 on a 28 day cycle.
  Other Names: Istodax

SUMMARY:
This is a study to test how safe the combination of the drugs Romidepsin and Pralatrexate are in patients with lymphoid malignancies and to determine the dose of the combination of drugs that is safest. If the combination is determined to be safe, the study will continue accrual patients with peripheral T-Cell lymphoma (PTCL).

DETAILED DESCRIPTION:
The non- Hodgkin lymphomas (NHL) represent a heterogeneous group of malignancies. Under the rubric of lymphoma exist some of the fastest growing cancers known to science, (Burkett's lymphoma, lymphoblastic lymphoma/leukemia), as well as some of the most indolent (small lymphocytic lymphoma, follicular lymphoma, and marginal zone lymphoma). This remarkable diversity of biology imposes significant challenges. Researchers are seeking to understand the cell of origin and differentiate what are sometimes subtle differences between the related sub-types of disease; and to identify the best treatments for these subtypes, with the ever-increasing likelihood that new understanding of the molecular pathogenesis of these diseases will result in an increase in new drugs for specific target populations.

ELIGIBILITY:
Inclusion Criteria:

Phase I: Patients must have histologically confirmed relapsed or refractory Non-Hodgkin's lymphoma, Hodgkin's Disease or multiple myeloma (defined by World Health Organization (WHO) criteria).

Phase II: Patients must have histologically confirmed relapsed or refractory T-Cell Lymphoma (as defined by WHO criteria).

* Must have received first line chemotherapy. No upper limit for the number of prior therapies
* Evaluable Disease
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patients must have adequate organ and marrow function as defined in the protocol
* Adequate Contraception
* Ability to understand and the willingness to sign a written informed consent document
* Inclusion Criteria for Multiple Myeloma patients specified in the protocol

Exclusion Criteria:

* Prior Therapy

  * Exposure to chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
  * Systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs
  * No other investigational agents are allowed
* Central nervous system metastases, including lymphomatous meningitis
* History of allergic reactions to Pralatrexate or Romidepsin
* Uncontrolled intercurrent illness
* Pregnant women
* Nursing women
* Current malignancy or history of a prior malignancy, as outlined in the protocol
* Patient known to be Human Immunodeficiency Virus (HIV)-positive
* Active Hepatitis A, Hepatitis B, or Hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of the combination of pralatrexate and romidepsin | Up to 1.5 years
  For Phase I
Overall response rate (ORR) (complete + partial response) of the combination of pralatrexate and romidepsin in patients with relapsed/refractory T-Cell Lymphoma | Up to 3 years
  For Phase II

SECONDARY OUTCOMES:
Maximum number of cycles received | Up to 1.5 years
  For Phase II
Number of dose delays at the MTD | Up to 1.5 years
  For Phase I
Overall response rate (ORR) of the study population | Up to 1.5 years
  For Phase I
Duration of response (DOR) of the combination in patients with T-Cell Lymphoma | Up to 3 years
  For Phase II
Overall survival (OS) of patients with T-Cell Lymphoma on study | Up to 3 years
  For Phase II
Progression free survival (PFS) of the combination in patients with T-Cell Lymphoma | Up to 3 years
  For Phase II
Number of dose reductions at the MTD | Up to 1.5 years
  For Phase I
Progression free survival (PFS) of the study population | Up to 1.5 years
  For Phase I
Duration of response (DOR) of the study population. | Up to 1.5 years
  For Phase I

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Amengual, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ryu Tiger YK, Jain S, Barta SK, Tolu S, Estrella B, Sawas A, Lue JK, Francescone MM, Pro B, Amengual JE. Phase II study of the novel antifolate agent pralatrexate in combination with the histone deacetylase inhibitor romidepsin for the treatment of patients with mature T-cell lymphoma. Leuk Lymphoma. 2024 Jun;65(6):736-745. doi: 10.1080/10428194.2024.2329996. Epub 2024 Mar 22. PMID 38517235
- [Derived] Amengual JE, Lichtenstein R, Lue J, Sawas A, Deng C, Lichtenstein E, Khan K, Atkins L, Rada A, Kim HA, Chiuzan C, Kalac M, Marchi E, Falchi L, Francescone MA, Schwartz L, Cremers S, O'Connor OA. A phase 1 study of romidepsin and pralatrexate reveals marked activity in relapsed and refractory T-cell lymphoma. Blood. 2018 Jan 25;131(4):397-407. doi: 10.1182/blood-2017-09-806737. Epub 2017 Nov 15. PMID 29141948